CLINICAL TRIAL: NCT01354145
Title: Twenty-four Month Exploratory Study of the Effect of Chondroitin Sulphate on Structural Changes in Knee Osteoarthritis Patients as Assessed by MRI
Brief Title: Study of the Effect of Chondroitin Sulfate on Structural Changes in Knee Osteoarthritis Patients Assessed by MRI
Acronym: MOSAIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS/III-DMOAD-02
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Chondroitin Sulfates; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chondroitin sulfate (Condrosan) (Experimental): CHONDROITIN SULPHATE Group: 1200 mg (three capsules of 400 mg each) taken once a day in the morning
  Interventions: Drug: Chondroitin sulfate
- Celecoxib (Active Comparator): CELECOXIB Group: 200 mg (one capsule of 200 mg CELECOXIB + two placebo capsules) taken in the morning
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Chondroitin sulfate — Chondroitin sulphate 1200 mg/day, 24 months treatment period
  Other Names: Condrosan
  Arms: Chondroitin sulfate (Condrosan)
Drug: Celecoxib — Celecoxib 200 mg/day, 24 months treatment period
  Arms: Celecoxib

SUMMARY:
The main purpose of this study is to compare the cartilage volume loss at the Baseline visit and after 24 months of treatment in patients treated with CHONDROITIN SULPHATE (CONDROSAN) 1200 mg daily vs. patients treated with CELECOXIB 200 mg daily.

DETAILED DESCRIPTION:
To compare long term disease modifiying and symptomatic effects at the Baseline visit and after 24 months of treatment in patients treated with CHONDROITIN SULPHATE 1200 mg daily vs. patients treated with CELECOXIB 200 mg daily.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of either sex, aged 40 years and more
* Subjects presenting primary OA of the knee according to ACR criteria with signs of synovitis (warmth, swelling or effusion
* OA of radiological stages 2 and 3 according to Kellgren-Lawrence;
* Minimum joint space width ≥2 mm in the medial femorotibial compartment on standing knee X-ray
* VAS of pain while walking ≥ 40 mm

Exclusion Criteria:

* Known allergy to CHONDROITIN SULPHATE, hypersensitivity to CELECOXIB, demonstrated allergic-type reactions to sulphonamides, experienced asthma, urticaria or allergic-type reactions after taking sulphonamides, aspirin (acetyl salicylic acid [ASA]), lactose or NSAIDs
* Active malignancy of any type or history of a malignancy within the last five years other than basal cell carcinoma
* Increased risk for prostate cancer, with prostate cancer, or with a history of prostate cancer within the last five years
* Subjects with other bone and articular diseases (antecedents and/or current signs) such as chondrocalcinosis, Paget's disease of the ipsilateral limb to the target knee, rheumatoid arthritis, aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, haemochromatosis, Wilson's disease, osteochondromatosis seronegative spondylo-arthropathy, mixed connective tissue disease, collagen vascular disease, psoriasis, inflammatory bowel disease
* Isolated knee lateral compartment OA defined by joint space loss in the lateral compartment only
* Class IV functional capacity using the American Rheumatism Association criteria
* Have had surgery in any lower limb or arthroscopy, aspiration or lavage in any lower limb joint within 180 days of the Baseline Visit
* History of heart attack or stroke, or experienced serious chest pain related to heart disease, or who have had serious diseases of the heart such as congestive heart failure
* High risk of CV events, according to the AHA assessment of CV risk tables
* History of recurrent UGI ulceration or active inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), a significant coagulation defect, or any other condition, which in the investigator's opinion might preclude the chronic use of CELECOXIB. Subjects may, at the Investigator's discretion, take a PPI or antacids daily as required
* Have been diagnosed as having or have been treated for oesophageal, gastric, pyloric channel, or duodenal ulceration within 30 days prior to receiving the first dose of study medication
* Subjects using corticosteroids (oral, injectable; exception of intraarticular/soft tissue injection at the exclusion of the target knee), indomethacin, tramadol, codeine, empracet, therapeutic dose of glucosamine or CHONDROITIN SULPHATE during the 12 weeks preceding inclusion
* Using hyaluronic acid (intra-articular target knee) during the 26 weeks preceding inclusion
* Using Natural Health Products (e.g. capsaicin, boswellia, willow bark), and creams and analgesic gels (e.g. camphor and alcohol based gels) during one week preceding baseline;
* Using Natural Health Products susceptible to increase the risk of bleeding (e.g. garlic, dong quai, etc.) during one week preceding baseline;
* Receiving radioactive synovectomy (target knee) during the 12 weeks preceding inclusion;
* Subjects who are receiving NSAID and do not want to stop during the study
* If treatment of osteoporosis (biphosphonates, SERMS, THS) is necessary, it will have to be continued, unmodified, for the entire duration of the study
* Have used medications with MMP-inhibitory properties (e.g. tetracycline or structurally related compounds) within 28 days prior to the Baseline Visit
* Are taking lithium carbonate, phenytoin or anticoagulants (with the exception of ASA up to a maximum daily dose of 325 mg)
* Have received chondrocyte transplants in any lower extremity joint
* Use oral or topical COXIBs, calcitonin or immunosuppressive drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2011-06; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Pelletier, MD, Study Chair — Principal Author
Locations (5):
- Canada (5):
  - Institut de Rhumatologie de Montréal, Montreal, Quebec
  - Osteoarthritis Research Unit, University of Montreal Hospital Research Centre (CRCHUM), Montreal, Quebec
  - Groupe de Recherche en rhumatologie et maladies osseoues, Québec, Quebec
  - Centre de Rhumatologie St. Louis, Sante Foi, Quebec
  - Centre de Recherche musculo-squellettique, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martel-Pelletier J, Raynauld JP, Mineau F, Abram F, Paiement P, Delorme P, Pelletier JP. Levels of serum biomarkers from a two-year multicentre trial are associated with treatment response on knee osteoarthritis cartilage loss as assessed by magnetic resonance imaging: an exploratory study. Arthritis Res Ther. 2017 Jul 20;19(1):169. doi: 10.1186/s13075-017-1377-y. PMID 28728606
- [Derived] Pelletier JP, Raynauld JP, Beaulieu AD, Bessette L, Morin F, de Brum-Fernandes AJ, Delorme P, Dorais M, Paiement P, Abram F, Martel-Pelletier J. Chondroitin sulfate efficacy versus celecoxib on knee osteoarthritis structural changes using magnetic resonance imaging: a 2-year multicentre exploratory study. Arthritis Res Ther. 2016 Nov 3;18(1):256. doi: 10.1186/s13075-016-1149-0. PMID 27809891

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib (Celebrex): CELECOXIB Group: 200 mg (one capsule of 200 mg CELECOXIB + two placebo capsules) taken in the morning
  Celecoxib: Celecoxib 200 mg/day, 24 months treatment period
Period: Overall Study
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Started | 97 | 97
Completed | 58 | 63
Not Completed | 39 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib | Total
Number analyzed (Participants) | 97 | 97 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 56 | 115
  >=65 years | 38 | 41 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (9.3) | 61.3 (8.5) | 61.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 36 | 80
  Male | 53 | 61 | 114
Cartilage Volume in the Lateral Compartment [Mean (Standard Deviation); unit: cubic milimeters] | 6606 (2332) | 6343 (1565) | 6475 (1985)
Cartilage Volume in the Medial Compartment [Mean (Standard Deviation); unit: cubic milimeters] | 6059 (2031) | 5705 (1572) | 5882 (1820)
Cartilage Volume in the Global Knee [Mean (Standard Deviation); unit: cubic milimeters] | 12665 (4259) | 12048 (2969) | 12356 (3674)

OUTCOME MEASURES:

1. Primary Outcome: Cartilage Volume Loss of the Lateral Compartment
Description: To compare the cartilage volume loss of the lateral compartment (femoral condyle and tibial plateau) at the Baseline visit and after 12 and 24 months of treatment either with CHONDROITIN SULPHATE (CONDROSAN) 1200 mg daily or with CELECOXIB 200 mg daily.
Time Frame: 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: cubic milimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
cubic milimeters
  Visit 6 (Day 364) | 6408 (97) | 6196 (97)
  Visit 9 (Day 728) | 6196 (99) | 6143 (99)

2. Secondary Outcome: Cartilage Volume Loss of the Global Knee
Description: To compare the cartilage volume loss of the global knee at the Baseline visit and after 12 and 24 months.
Time Frame: 12 months (Day 364) and 24 months (Day 728)
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: cubic milimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
cubic milimeters
  Visit 6 (Day 364) | 12210 (175) | 11770 (175)
  Visit 9 (Day 728) | 11877 (179) | 11572 (179)

3. Secondary Outcome: Cartilage Volume in the Medial Compartment
Description: To compare the cartilage volume loss of the medial compartment at the Baseline visit and after 12 and 24 months.
Time Frame: 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: cubic milimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
cubic milimeters
  Visit 6 (Day 364) | 5793 (83) | 5586 (84)
  Visit 9 (Day 728) | 5672 (87) | 5439 (87)

4. Secondary Outcome: Synovial Membrane Thickness
Description: To compare the severity of synovitis score (Thickness of the Synovial Membrane in mm) in Global Knee , at the baseline visit and the follow-up visits in subjects treated either with CHONDROITIN SULPHATE (CONDROSAN) or CELECOXIB.
  The severity of synovitis was evaluated through four regions of interest (ROIs) in the images of the axial T1-weighted acquisition complemented with the use of the images of the axial T2-weighted acquisition. The thickness of the synovial membrane was evaluated in the global knee and each of the ROIs and results were expressed in millimetres. The four ROIs were the proximal lateral, distal lateral, proximal medial and distal medial.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
milimeters
  Visit 2 (Baseline) | 0.99 (0.22) | 0.96 (0.22)
  Visit 6 (Day 364) | 1.05 (0.22) | 1.07 (0.26)
  Visit 9 (Day 728) | 1.19 (0.26) | 1.16 (0.31)

5. Secondary Outcome: Bone Marrow Lesions Score
Description: To compare the bone marrow lesions (BMLs) score in the global knee and the different sub regions at the baseline visit and the follow-up visits in subjects treated either with CHONDROITIN SULPHATE (CONDROSAN) or CELECOXIB.
  The BMLs were assessed in the global knee and the different sub region of the knee (medial trochlea, plateau of the medial femoro-tibial joint, femur of the medial femoro-tibial joint, medial posterior condyle, lateral trochlea, plateau of the lateral femoro-tibial joint, femur of the lateral femoro-tibial joint, lateral posterior femur). The BMLs score was defined as a grade (between 0 and 3) in each knee sub region and summed to derive a global knee score ranging between 0 (absent) and 30 (present). Specifically, each grade was scored as follows:
  * Grade 0 = Absence of lesion in the sub region
  * Grade 1 = less than 25% of the surface
  * Grade 2 = 25-50% of the surface
  * Grade 3 = more than 50% of the surface
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
units on a scale
  Global Knee - Visit 2 (Baseline) | 2.57 (3.04) | 2.65 (2.51)
  Global Knee - Visit 6 (Day 364) | 3.16 (3.53) | 2.77 (2.40)
  Global Knee - Visit 9 (Day 728) | 3.58 (3.68) | 3.37 (2.83)

6. Secondary Outcome: Synovial Fluid Volume
Description: To compare the synovial fluid volume of the global knee at the Baseline visit and after 24 months.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: mililiters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
mililiters
  Visit 2 (Baseline) | 13.83 (14.61) | 10.79 (10.94)
  Visit 6 (Day 364) | 10.30 (10.08) | 9.49 (12.06)
  Visit 9 (Day 728) | 10.97 (14.52) | 9.07 (13.60)

7. Secondary Outcome: Percentage of Participants With the Presence of Extrusion in the Meniscus
Description: The presence of a meniscal extrusion was assessed in each of sub regions. The absence of a severe extrusion in all the sub regions was considered as an absence (score=0) of a severe extrusion in the meniscus. The presence of a severe extrusion in at least one region of the meniscus was sufficient to consider the presence (score=1) of a severe extrusion in the meniscus.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Number; unit: percentage of participants
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
percentage of participants
  Visit 2 (Baseline) Medial meniscus | 47.4 | 47.4
  Visit 6 (Day 364) Medial meniscus | 53.6 | 53.6
  Visit 9 (Day 728) Medial meniscus | 56.1 | 60.3
  Visit 2 (Baseline) Lateral meniscus | 6.2 | 3.1
  Visit 6 (Day 364) Lateral meniscus | 7.2 | 2.9
  Visit 9 (Day 728) Lateral meniscus | 8.8 | 3.2

8. Secondary Outcome: Visual Analog Scale (VAS)
Description: Visual Analogue Scale: 0 No Pain 10 Maximum Pain Huskisson's VAS measures global pain intensity. Patients were asked to quantify their disease status on a 10 cm VAS as follows: "Please indicate the severity of knee pain experienced during the last 48 hours by marking a (I) through the line". Left hand marker represents "No pain" and right hand marker represents "The worst pain imaginable".
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
centimeters
  Visit 2 (Baseline) | 6.24 (1.55) | 5.93 (1.81)
  Visit 6 (Day 364) | 3.43 (2.60) | 3.02 (2.51)
  Visit 9 (Day 728) | 3.12 (2.85) | 2.45 (2.33)

9. Secondary Outcome: WOMAC Pain Subscale
Description: Western Ontario & McMaster Universities Osteoarthritis Index (WOMAC) Pain subscale Score Range: 0 (no pain) - 50 (maximum pain) The study was designed such that the outcome of primary interest is knee pain related to OA. The measure selected to best evaluate this is an improvement in the WOMAC pain subscales. This subscale consists of 5 items which assesses the pain during walking, using stairs, in bed, sitting or lying, and standing.Each item is a 10 cm VAS with 0 and 10 cm representing no pain and extreme pain respectively.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
centimeters
  Visit 2 (Baseline) | 25.6 (8.11) | 25.51 (9.04)
  Visit 6 (Day 364) | 14.71 (11.55) | 13.62 (11.49)
  Visit 9 (Day 728) | 13.51 (12.67) | 10.69 (10.66)

10. Secondary Outcome: WOMAC Stiffness Subscale
Description: Western Ontario & McMaster Universities Osteoarthritis Index, from 0 No Stiffness to 20 Maximum Stiffness WOMAC stiffness subscale was used to measure the stiffness of the knee with pain. Two items are used to assess stiffness grade: after first waking and later in the day.Each item is a 10 cm VAS with 0 and 10 cm representing no difficulty and extreme difficulty respectively.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
centimeters
  Visit 2 (Baseline) | 10.76 (3.68) | 11.65 (4.25)
  Visit 6 (Day 364) | 6.53 (4.76) | 6.60 (5.31)
  Visit 9 (Day 728) | 6.15 (5.27) | 5.44 (5.28)

11. Secondary Outcome: WOMAC Function Subscale
Description: Western Ontario & McMaster Universities Osteoarthritis Index, from 0 No Function to 170 Maximum Function WOMAC functional limitation subscale was used to measure the functionality of the knee with pain. Seventeen items are used to assess functionality of the knee: tair use, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy household duties, light household duties. Each item is a 10 cm VAS with 0 and 10 cm representing no difficulty and extreme difficulty respectively.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
centimeters
  Visit 2 (Baseline) | 88.5 (28.7) | 89.5 (32.5)
  Visit 6 (Day 364) | 52.3 (39.1) | 51.0 (42.7)
  Visit 9 (Day 728) | 50.0 (44.4) | 46.2 (41.4)

12. Secondary Outcome: Short Form (SF-36) Health Survey
Description: The SF-36 is composed of 35 items measuring:
  * 8 health concepts (or dimensions), [(Physical Functioning (PF), Role Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE) and Mental Health (MH)]
  * and 1 reported health transition item.
  The 8 health concepts are summarized in 1 physical (PCS) and 1 mental (MCS) component summary measures. PCS is represented by physical function, role limitations-physical, pain, and general health perception. MCS is represented by vitality, social function, role limitations-emotional, and mental health. Subscale items are summed and scaled from 0-100 to give subscale scores; 0= worst health related quality of life (HRQL), 100=best HRQL. PCS and MCS summary scores are constructed as T-scores (mean =50, standard deviation=10) with no minimum or maximum score; higher scores indicate better health status.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Median (Standard Deviation); unit: Scores on a scales
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
Scores on a scales
  Visit 2 (Baseline) Physical Component Summary | 35.4 (7.8) | 35.7 (8.1)
  Visit 6 (Day 364) Physical Component Summary | 39.6 (9.6) | 41.6 (10.1)
  Visit 9 (Day 728) Physical Component Summary | 41.8 (9.5) | 42.2 (10.0)
  Visit 2 (Baseline) Mental Component Summary | 51.7 (9.5) | 52.7 (11.0)
  Visit 6 (Day 364) Mental Component Summary | 53.2 (9.0) | 54.0 (10.7)
  Visit 9 (Day 728) Mental Component Summary | 52.7 (9.2) | 56.0 (8.0)

13. Secondary Outcome: Percentage of Participants With Presence of Joint Swelling and Effusion
Description: Study knees were evaluated at each visit for the presence or absence of swelling and effusion.
Time Frame: Baseline, 12 months (Day 364) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Number; unit: percentage of participants
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
percentage of participants
  Baseline | 60.8 | 56.7
  Visit 9 (Day 728) | 10.3 | 17.7

14. Secondary Outcome: Use of Acetaminophen
Description: Consumption of Acetaminophen: At each post-baseline visit, the investigator had to assess the consumption of acetaminophen, rescue analgesic authorised throughout the study, by reporting the number of caplets dispensed/retrieved since the previous visit.
  Daily consumption of acetaminophen was calculated as an average.
Time Frame: 3 months (Day 91), 6 momnths (Day 182), 12 months (Day 364), 18 monts (Day 546) and 24 months (Day 728)
Population: Intention-To-Treat
Measure: Mean (Standard Deviation); unit: Daily number of caplets taken
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib (Celebrex)
Number analyzed (Participants) | 97 | 97
Daily number of caplets taken | 1.17 (1.43) | 0.94 (1.61)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Chondroitin Sulfate (Condrosan) | Celecoxib
Serious Adverse Events (participants affected / at risk) | 10/97 | 6/97
Other Adverse Events (participants affected / at risk) | 78/97 | 79/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chondroitin Sulfate (Condrosan) (N=97) | Celecoxib (N=97)
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 0 | 1
Morganella Infection (Infections and infestations) | 1 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip And/Or Oral Cavity Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cataract Operation (Surgical and medical procedures) | 1 | 0
Hip Surgery (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Diverticular Perforation (Gastrointestinal disorders) | 0 | 1
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Proctocolitis (Gastrointestinal disorders) | 1 | 0
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 1 | 0
Urinary Retention Postoperative (Injury, poisoning and procedural complications) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Sinus Arrhythmia (Cardiac disorders) | 1 | 0
Bladder Perforation (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chondroitin Sulfate (Condrosan) (N=97) | Celecoxib (N=97)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 17 | 5
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 8
Nasopharyngitis (Infections and infestations) | 28 | 18
Dyspepsia (Gastrointestinal disorders) | 12 | 12
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 5 | 5
Headache (Nervous system disorders) | 15 | 10
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 18 | 18
General disorders and administration site conditions (General disorders) | 12 | 12
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 3 | 11
Psychiatric disorders (Psychiatric disorders) | 4 | 9
Investigations (Investigations) | 6 | 6
Surgical and medical procedures (Surgical and medical procedures) | 8 | 8
Vascular disorders (Vascular disorders) | 7 | 5
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 30 | 32
Infections and infestations (Infections and infestations) | 38 | 43
Gastrointestinal disorders (Gastrointestinal disorders) | 20 | 27
Nervous system disorders (Nervous system disorders) | 6 | 12
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 14 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less